CLINICAL TRIAL: NCT04258085
Title: Promoting Earlier Detection of Breast Cancer in Rwanda: Scaleup in the National Health Care System
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Rwanda Biomedical Centre (Other); Partners in Health (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Lydia Pace, MD, MPH, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2014P002688a
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Benign Breast Disease
Keywords: Rwanda; breast cancer; screening; early detection
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening plus EMR: Individuals in this group are those residing in districts where health facilities have implemented a breast cancer screening program integrated with cervical cancer screening, the Women's Cancer Early Detection Program (WCEDP).
  Interventions: Other: Early diagnosis program combined with electronic medical record

INTERVENTIONS:
Other: Early diagnosis program combined with electronic medical record — Implementation of early diagnosis approach targeting symptomatic women, combined with use of electronic medical record to facilitate documentation, patient tracking across levels of the health care system, and patient contact

SUMMARY:
This observational study evaluates scale-up of a breast cancer early detection program in Rwanda that was initially piloted in a single district. Specifically investigators will examine patient volume, service delivery, loss-to-follow-up rates, and cancer detection rates noted following implementation of scale-up to 3 additional districts. For scaleup, breast cancer screening with CBE was added to a cervical cancer screening initiative, in a combined Women's Cancer Early Detection Program (WCEDP).

DETAILED DESCRIPTION:
Investigators previously conducted a cluster randomized controlled trial of a clinician training program to facilitate prompt evaluation of women with breast symptoms in one rural district of Rwanda. Subsequently, Rwanda Biomedical Centre (RBC) has scaled up the curriculum in 3 districts, adapting the program to integrate CBE screening into a cervical cancer screening initiative. In this study, we will evaluate implementation of this combined screening initiative. Investigators will assess patient volume, services, diagnoses, and loss to follow up.

ELIGIBILITY:
Inclusion Criteria:

* All women and men who are evaluated for a breast concern or receive breast cancer screening through implementation of the nationally-led early detection programs

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is the population served by the health centers that are implementing the nationally-led breast cancer early detection program.
Sampling Method: Non-Probability Sample
Enrollment: 17379 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Cancer detection rate | 2 years
  Proportion of patients presenting to health centers who are ultimately diagnosed with cancer; proportion of patients who receive biopsy who are ultimately diagnosed with cancer; proportion of individuals diagnosed with cancer who initially presented with versus without breast symptoms
Loss to follow-up | one year
  Rates of loss-to-follow up before and after implementation of electronic medical record in districts utilizing breast cancer screening approach; and loss to follow up in districts implementing early diagnosis approach and EMR
Patient volume and services received | two years
  Number of patients presenting at the health centers, district hospital and referral hospitals

SECONDARY OUTCOMES:
Breast cancer stage | 2 years
  Among women diagnosed with breast cancer, distribution of cancer stage among women who participated in the WCEDP.
Patients' costs | 6 months
  out-of-pocket costs borne by patients while undergoing evaluation for an abnormal clinical breast exam

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Pace, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Rwanda Biomedical Centre, Kigali, Rwanda